CLINICAL TRIAL: NCT00925418
Title: Randomized Trial Evaluating the Cryotherapy in the Prevention of Nails Toxicity Induced by Taxotere® in Patient Treated for Breast or Prostate Cancer.
Brief Title: Evaluation of the Cryotherapy in the Prevention of Nails Toxicity Induced by Taxotere® in Breast or Prostate Cancer
Acronym: CRYO1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRYO 1/IPC 2005-007
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Breast Neoplasms; Prostate Cancer; Nail Diseases
Keywords: Neoplasm; breast Neoplasm; docetaxel; Glove
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Nail Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without Glove (No Intervention): Patients do not use frozen glove during chemotherapy with Taxotere®
- With Glove (Experimental): Patients use frozen glove during chemotherapy with Taxotere®
  Interventions: Procedure: Frozen Glove

INTERVENTIONS:
Procedure: Frozen Glove — Using frozen glove during chemotherapy with Taxotere®
  Arms: With Glove

SUMMARY:
Taxotere® can induce nails changes like dyschromia, hematoma, lines of Beau-Reil (signing the stop of the epithelial proliferation), abscess, or pain. In this context, this randomized, monocentric phase III trial evaluates the cryotherapy, using frozen glove, in the prevention of nails toxicity induced by Taxotere® in patient treated for breast or prostate cancer.

Primary objective:

Demonstrate a reduction of the nails toxicity using frozen glove during chemotherapy with Taxotere®.

Secondary objectives:

Analysis of time of protection against onycholysis Estimation of the efficiency of cryotherapy, and impact on quality of life Tolerance and compliance of the frozen glove

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormono-resistant breast cancer or metastatic prostate cancer treated by chemotherapy with Taxotere®.
* Patients aged 18 and older
* Nail toxicity < grade 2 (CTC-AE version 3.0)
* Informed patients with signed consent

Exclusion Criteria:

* History of treatment with taxane
* Raynaud syndrome
* Distal metastasis in superior extremity
* Nail diseases
* Distal arteriopathy
* Cold intolerance
* Peripheral neuropathy>=2
* Pregnancy, breast feeding
* Unable to give informed consent
* Unable to have a medical follow-up for social, geographical, family or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of patients treated by Taxotere® with nail toxicity >= 2 (CTC-AE version 3.0) | 4 months

SECONDARY OUTCOMES:
Number of day between inclusion and apparition of nail toxicity | 4 months
Necessity of local care, existence of pains | 4 months
Tolerance and compliance for the frozen glove | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carole TARPIN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut PAOLI-CALMETTES, Marseille, France

REFERENCES:
- See also: Official web site of the sponsor — http://www.institutpaolicalmettes.fr